CLINICAL TRIAL: NCT02617212
Title: Impact of Implant Abutment Dis-/Reconnection on Peri-Implant Marginal Bone Loss - Randomized Clinical Trial.
Brief Title: Implant Abutment Dis-/Reconnection and Peri-Implant Marginal Bone Loss.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Collaborators: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Luciano de Freitas Guimarães Praça, MS, Fortaleza University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.310.562
Record Dates: First submitted 2015-11-19; First posted 2015-11-30 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Alveolar Bone Loss
Keywords: dental implant; bone preservation; definitive abutment; one abutment one time
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Definitive abutment (Experimental): Implant surgery. No abutment dis-/reconnections.
  Interventions: Procedure: Implant surgery; Device: No abutment dis-/reconnections.
- Conventional treatment (Active Comparator): Implant surgery. Three abutment dis-/reconnections.
  Interventions: Procedure: Implant surgery; Device: Three abutment dis-/reconnections.

INTERVENTIONS:
Procedure: Implant surgery — The volunteers will receive one or two dental implant(s) placed by a surgical procedure, under local anesthesia and careful soft and hard tissue handling. After implant insertion, the volunteers will be randomly assigned to one arm.
Device: Three abutment dis-/reconnections. — At the active comparator arm, each implant will receive a titanium healing abutment during the surgery, according to manufacturer's recommendations. Three dis-/reconnections of abutments will be performed after the soft tissue healing period: the first, after 8 weeks, for adjustment of the emergence profile by healing abutment changing; the second, 10 weeks after surgery, for intra-oral prosthetic abutment selection; and the third, 12 weeks after surgery, for the prosthetic abutment definitive connection with the manufacturer recommended torque.
  Arms: Conventional treatment
Device: No abutment dis-/reconnections. — Each experimental arm implant will receive its definitive prosthetic abutment at the surgical procedure. The manufacturer recommended torque will be applied so that no disconnection of the abutment will occur during and after completion of the treatment. The abutment will receive healing caps, which shall remain in position until the end of 12 weeks after surgery.
  Arms: Definitive abutment

SUMMARY:
The purpose of this study is to investigate whether the immediate definitive abutment connection to dental implant is effective in preventing marginal bone loss when compared to the conventional treatment with late abutment/implant connection, which include three disconnections and reconnections.

DETAILED DESCRIPTION:
The proposed study is a randomized clinical trial in which the participants will be allocated into one of the two arms according to the proposed intervention: experimental group, in which the abutments will be permanently connected immediately at the implant placement procedure; and control group (active comparator) with conventional treatment, where the abutments will be disconnected and reconnected three times.

Considering the inclusion and exclusion criteria related to oral and systemic health, a sample of participants will be selected among those partially edentulous patients who seek for dental implants treatment at the Fortaleza University School of Dentistry.

The sample size has been calculated based on the standard deviation of 0.17 mm, significance level of 5% and 80% statistical test power. To detect a clinically significant difference of 0.2 mm, each group should be composed of 11 participants. Therefore, considering a 10% margin for possible dropouts or missing data, the study will include 24 participants divided into two groups. Each participant will receive one or two implants according to his/her needs, so the study may include more than 24 implants.

A single surgeon will perform the implant surgical procedure in order to reduce variations inherent to clinical experience. After local anesthesia and incision on the top of the alveolar ridge, the bone will be exposed by the mucoperiosteal flap elevation. The mucosal thickness will be measured at implant sites, before the lingual/palatal flap elevation, with a periodontal probe.

The drilling sequence will be done according to manufacturer's recommendations, under saline solution irrigation, intermittent movements and speed up to 1200rpm.

The implants should develop a final insertion torque of 32Ncm or above to enable abutment connection torque, indicated at the experimental arm. The implant primary stability will be also measured by resonance frequency analysis (Osstell; Osstell AB, Gothenburg, Sweden). A minimum 65 ISQ will be required to a single-stage surgery. Thus, those implants that do not contemplate these requirements will be excluded from the study and will receive a conventional treatment with two-stage surgery if necessary.

Before finishing the surgical procedure, the volunteers will be randomly assigned to one of the two arms by opening sealed envelopes with a random sequence generated by Excel (Microsoft, Redmond, Washington, USA). Therefore, the surgeon will identify each volunteer's arm only after the end of drilling, insertion and stabilization of the implants.

Each implant allocated at the control arm (active comparator) will receive conventional treatment with three abutment disconnections and reconnections. At the experimental arm, each implant will receive the prosthetic abutment in a definitive way immediately at the surgical procedure, avoiding any abutment disconnection.

The surgeries of both arms will be finished with suture, drug prescription and postoperative recommendations. All implants will receive temporary crowns at three months and definitive prosthesis until six months after surgery.

Intraoral radiographs will be done with paralleling technique immediately after surgery (baseline) and at 3, 6, 12 and 24 months later. The radiographs will have its dimensions corrected at the ImageJ software (National Institutes of Health, Bethesda, Maryland, USA) having implant known dimensions as reference.

Each implant will have its radiographs evaluated by a previously calibrated examiner with a minimum of 0.8 intra-rater reliability for the intraclass correlation coefficient. The examiner will not know to which arm the X-rays belong.

Primary and secondary outcomes data will be submitted to normality test and compared using statistical tests for paired and unpaired samples.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients requiring dental implant treatment for one or two dental units;
* Occlusal stability and regular occlusal plane;
* Enough space for implant and prosthesis;
* Good periodontal health
* Keratinized mucosa width > 4mm;
* Implant primary stability > 65 ISQ and insertion torque > 20Ncm;

Exclusion Criteria:

* Diabetes mellitus;
* Treatment with bisphosphonates;
* Head and neck irradiation;
* General contraindications to oral surgery;
* Pregnancy;
* Bone graft;
* Bruxism;
* Smoking habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Peri-implant marginal bone level change. | 2, 6, 12 and 24 months after implant surgery.
  To estimate the gingival margin stability and the long-term success of implant-supported restorations, the peri-implant marginal bone level will be assessed as primary outcome through intraoral radiographs, in a perspective of bone maintenance, bone loss or bone gain.

SECONDARY OUTCOMES:
Implant stability change. | 3 and 6 months after implant surgery.
  The implant stability will be measured using a resonance frequency analysis equipment to confirm the implant osseointegration.
Gingival level change. | 6, 12 and 24 months after implant surgery.
  The gingival level will be measured using a periodontal probe and an acrylic stent as a reference.
Peri-implant probing depth change. | 12 and 24 months after implant surgery.
  To evaluate the peri-implant health, the probing depth will be assessed in 6 areas around the implant using the prosthetic abutment as a reference.
Bleeding on probing change. | 12 and 24 months after implant surgery.
  To evaluate the peri-implant health, the bleeding on probing will be observer or not at until 10 seconds after peri-implant probing.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo O. Rego, PhD, Study Director — Universidade Federal do Ceara
Locations (1):
- Fortaleza University; Health Sciences Center; School of Dentistry., Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Abrahamsson I, Berglundh T, Lindhe J. The mucosal barrier following abutment dis/reconnection. An experimental study in dogs. J Clin Periodontol. 1997 Aug;24(8):568-72. doi: 10.1111/j.1600-051x.1997.tb00230.x. PMID 9266344
- [Background] Tarnow DP, Cho SC, Wallace SS. The effect of inter-implant distance on the height of inter-implant bone crest. J Periodontol. 2000 Apr;71(4):546-9. doi: 10.1902/jop.2000.71.4.546. PMID 10807116
- [Background] Lazzara RJ, Porter SS. Platform switching: a new concept in implant dentistry for controlling postrestorative crestal bone levels. Int J Periodontics Restorative Dent. 2006 Feb;26(1):9-17. PMID 16515092
- [Background] Canullo L, Bignozzi I, Cocchetto R, Cristalli MP, Iannello G. Immediate positioning of a definitive abutment versus repeated abutment replacements in post-extractive implants: 3-year follow-up of a randomised multicentre clinical trial. Eur J Oral Implantol. 2010 Winter;3(4):285-96. PMID 21180681
- [Background] Pieri F, Aldini NN, Marchetti C, Corinaldesi G. Influence of implant-abutment interface design on bone and soft tissue levels around immediately placed and restored single-tooth implants: a randomized controlled clinical trial. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):169-78. PMID 21365053
- [Background] Becker K, Mihatovic I, Golubovic V, Schwarz F. Impact of abutment material and dis-/re-connection on soft and hard tissue changes at implants with platform-switching. J Clin Periodontol. 2012 Aug;39(8):774-80. doi: 10.1111/j.1600-051X.2012.01911.x. Epub 2012 Jun 7. PMID 22676071
- [Background] Rodriguez X, Vela X, Mendez V, Segala M, Calvo-Guirado JL, Tarnow DP. The effect of abutment dis/reconnections on peri-implant bone resorption: a radiologic study of platform-switched and non-platform-switched implants placed in animals. Clin Oral Implants Res. 2013 Mar;24(3):305-11. doi: 10.1111/j.1600-0501.2011.02317.x. Epub 2011 Oct 3. PMID 22092773
- [Background] Iglhaut G, Becker K, Golubovic V, Schliephake H, Mihatovic I. The impact of dis-/reconnection of laser microgrooved and machined implant abutments on soft- and hard-tissue healing. Clin Oral Implants Res. 2013 Apr;24(4):391-7. doi: 10.1111/clr.12040. Epub 2012 Sep 26. PMID 23009248